CLINICAL TRIAL: NCT01587976
Title: Health Related Quality of Life After Surgery and Oncological Treatment of Colorectal Liver Metastases A Prospective Multicenter Study
Brief Title: Health Related Quality of Life After Surgery and Oncological Treatment of Colorectal Liver Metastases
Acronym: HQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011/570
Record Dates: First submitted 2012-02-27; First posted 2012-04-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2013-09

CONDITIONS: Metastasis; Quality of Life
Keywords: Health related quality of life; Colorectal liver metastasis; surveillance
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to study health related quality of life (HQoL)after resection of colorectal liver metastases combined with perioperative chemotherapy. The investigators want to study if an aggressive, life prolonging and multimodal treatment can be defended from a quality of life perspective.

DETAILED DESCRIPTION:
Background: Hepatic resection is the only treatment with potential curative intent for patients having colorectal liver metastases. Combined with chemotherapy, the overall 5-year survival is 40-50%. The disease free 5-year survival is about 20%, and about 70% of resected patients experience recurrence from their disease. Even if surgery is superior all other treatments, most patients will finally die from their cancer. However; surgery contributes by adding years of life, and for a minority, a disease free life. There has been much effort to study predictors for outcome after surgery, but little has been focused on quality of life following this treatment.

Method: EORTC Validated questionnaire (European Organisation Research of Treatment of Cancer) version QLQ-C30 (3.0) and QLQ LMC21. The patients fill out the questionnaire before surgery as a baseline, and then after 3,6 and 12 months after surgery. The investigators also register important clinicopathological data about each patient prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Liver metastasis from colorectal cancer
* Resectability, with intension of R0 resection
* No macroscopic tumor left after surgery
* Patients with combined resectable extrahepatic tumors are also included.
* Patients must complete the questionnaire before the operation.

Exclusion Criteria:

* Drop out of questionnaire after surgery
* Patients found to be irresectable during the operation or where macroscopic tumor tissue are left behind.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with resectable colorectal liver metastases treated at Haukeland and Stavanger University hospital, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life after liver resection in combination with chemotherapy | 12 months after surgery
  The EORTC board has made validated questionaries with manuals for measuring quality of life. The important focus is to see if and when patients gain their HQoL as they did have before surgery.

SECONDARY OUTCOMES:
Identifying possible clinical parameters influencing the HQoL after liver resection. | Up to one year after surgery, maybe longer
  Examples of parameters: complications, extent of surgery, chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: August Bakke, Professor, Study Director — Director, Surgical clinic, Haukeland University Hospital, Helse-Bergen HF, N-5020 Bergen, Norway
Locations (1):
- Departement of acute and digestive surgery, surgical clinic, Haukeland University Hospital, Bergen, Bergen, Norway